CLINICAL TRIAL: NCT00263120
Title: Effects of Thymectomy During Cardiothoracic Surgery
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Nancy Halnon, MD, MS, Principal Investigator, University of California, Los Angeles
Other Study IDs: 2005-12-003Halnon
Record Dates: First submitted 2005-12-05; First posted 2005-12-07 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Thymectomy and Cardiothoracic Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Pain Questionnaire

SUMMARY:
The thymus is known to be the site of T cell development in humans. Due to its location in the chest in front of the heart, incidental thymecomy is commonly performed during cardiothoracic surgery, especially in infants and children, so that surgeons may gain access to the surgical field. This practice has been considered safe because it was thought that the thymus is inactive after birth. However, recent data using newly developed techniques has demonstrated that the thymus normally is active well into adulthood. In addition, in a previous study (UCLA IRB # 02-03-008-02) we have demonstrated alterations in lymphocyte (T cells) number in individuals who have undergone thymectomy in childhood but we do not know how immunity is affected. We plan to investigate if immune development or immune function later in life is affected by the loss of T cell production caused by thymectomy during cardiothoracic surgical procedures in childhood. At UCLA, a large number of patients are seen who have congenital heart disease and undergo surgical procedures for correction or repair and many children and adults are followed for many years after they have undergone surgical procedures. Subjects for study will be recruited from among these patients.

We propose a study which will examine the number and activity of lymphocytes obtained from blood samples from child and young adult subjects who have undergone surgery in early childhood. We will determine if these subjects have had complete thymectomy in the past using CT or MRI (obtained during routine care) or, for subjects who are having cardiothoracic surgery, by visualization of thymic tissue during the procedure. In addition we will give vaccination for a common viral illness (hepatitis A) and measure immune responses to it (from a blood sample). As part of this study, we will ask for medical information consisting of a history of congenital cardiac disease and other diagnoses (such as asthma), a history of infections and hospitalizations, and information about immunizations. We will also ask about a list of specific symptoms which will give us information about the function of the immune system.

ELIGIBILITY:
Inclusion Criteria:

* Age: birth to 35 years.
* Planning cardiac surgical procedure at UCLA Medical Center.
* For subjects with a history of prior cardiothoracic surgery: undergoing CT or MRI evaluation prior to reoperation.

Exclusion Criteria:

* Unable to travel to UCLA Medical Center for follow up blood tests (infants and young children in longitudinal study)
* Known thymus/immune deficiency disorder (i.e. DiGeorge Syndrome)

Max Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: child and young adult subjects who have undergone surgery in early childhood for correction or repair related to congenital heart disease enrolled for the observational portion of this protocol only
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2006-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
immune dysfunction | late

CONTACTS AND LOCATIONS:
Overall Officials: Nancy J. Halnon, M.D., Principal Investigator — Pediatric Cardiology, UCLA
Locations (1):
- UCLA Adult Congenital Heart Disease Clinic, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Halnon NJ, Jamieson B, Plunkett M, Kitchen CM, Pham T, Krogstad P. Thymic function and impaired maintenance of peripheral T cell populations in children with congenital heart disease and surgical thymectomy. Pediatr Res. 2005 Jan;57(1):42-8. doi: 10.1203/01.PDR.0000147735.19342.DE. Epub 2004 Nov 5. PMID 15531736
- [Result] Halnon NJ, Cooper P, Chen DY, Boechat MI, Uittenbogaart CH. Immune dysregulation after cardiothoracic surgery and incidental thymectomy: maintenance of regulatory T cells despite impaired thymopoiesis. Clin Dev Immunol. 2011;2011:915864. doi: 10.1155/2011/915864. Epub 2011 Jul 6. PMID 21776289